CLINICAL TRIAL: NCT06522802
Title: Does Wearing a Mask Affect Balance and Reaction Time?
Brief Title: The Effect of Wearing a Mask for Balance and Reaction Time
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, yasin yildirim, Physiotherapist, MSc, PhD, Istanbul Medipol University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 10840098-772.02-E.43565
Record Dates: First submitted 2024-07-12; First posted 2024-07-26 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Reaction Time; Balance

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Evaluation Arm (Experimental): Only one group evaluated
  Interventions: Diagnostic Test: balance tests, reaction time evaluation

INTERVENTIONS:
Diagnostic Test: balance tests, reaction time evaluation — Only 3 tests were applied to participants

SUMMARY:
A mask is a protective equipment that covers the mouth and nose and is routinely used in workplaces, public transport and other communal settings preventing harmful particles, dust, droplets, bacteria, viruses, fog, gas, smoke and steam from entering the respiratory system. However, wearing a mask may impair the visual field, potentially affecting balance and reaction time. The investigators' aim is to determine whether the use of masks affects people's balance and reactions.

ELIGIBILITY:
Inclusion Criteria:

* To be healthy

Exclusion Criteria:

* present or previous balance disorder

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2020-12-08 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2022-01-10 (Actual)

PRIMARY OUTCOMES:
Functional reach test | baseline-5 hours later
  Functional Reach Test (FRT) is a clinical outcome measure and assessment tool for ascertaining dynamic balance in in simple task. As we know that this test measures the distance between the length of an outstretched arm in a maximal forward reach, while maintaining a fixed base of support.

SECONDARY OUTCOMES:
COP displacement | baseline-5 hours later
  Displacement of the center of pressure (COP) and center of gravity (COG) a: COP ML displacement. Distance of the inflection point from a stationary baseline. b: Maximum ML separation. Maximum distance between the COP and COG. Source publication.
BlazePod evaluation | baseline-5 hours later
  A new technology (BlazePod™) that measures response time (RT) is currently on the market and has been used by strength and conditioning professionals.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University, Istanbul, Beykoz, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No